CLINICAL TRIAL: NCT06116175
Title: Efficacy of Continuous Radiofrequency 60 Celsius Degree in Management of Chronic Lateral Epicondylitis Prospective Study
Brief Title: Lateral Epicondylitis Continuous Radiofrequency Microtenotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iraqi Board of medical specialties (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M mahdi pain clinic
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- lateral epicondylitis (Experimental): chronic patients of tennis elbow
  Interventions: Procedure: 60 degree thermal radiofequency of tennis elbow

INTERVENTIONS:
Procedure: 60 degree thermal radiofequency of tennis elbow — under strict aseptic technique ultrasound guided TRF of lateral epicondylitis advanced for 5 mm active tip canula

SUMMARY:
prospective study measuring the outcome of continuous radio frequency 60 degree on lateral epicondylitis not responding to traditional ultrasound guided injection

ELIGIBILITY:
Inclusion Criteria:

* chronic tennis elbow no response to traditional injection ultrasound exam reveal swelling of common extensor tendon

Exclusion Criteria:

* complete tear of common extensor tendon implanted pace maker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
decrease in pain score after CRF | 6 months
  decrease in numerical analogue score

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
prospective study measuring the outcome of CRF in tennis elbow